CLINICAL TRIAL: NCT06400953
Title: The Effect of Kinetic Brain Exercises on Balance and Dual Task Activities in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Arzu Razak Ozdinçler, Head of department, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Brain Exercises in the Elderly
Record Dates: First submitted 2024-04-28; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Elderly; Exercise
Keywords: Kinetic Brain Exercises; Balance; Dual Task Performance; Elderly; Core Stabilization
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Kinetic Brain Exercises and Core Stabilization Exercises were applied to Group 1
  Interventions: Other: Kinetic Brain Exercises and Core Stabilization Exercises; Other: Core Stabilization Exercises
- Group 2 (Experimental): Core Stabilization Exercises were applied to Group 2
  Interventions: Other: Core Stabilization Exercises

INTERVENTIONS:
Other: Kinetic Brain Exercises and Core Stabilization Exercises — Kinetic Brain Exercise Program Kinetic brain exercises were applied to Group 1 in groups of 8-10 people, 2 days a week for 40 minutes for 8 weeks.These exercises include warm-up, main and cool-down phases. Warm-up; These are coordination-oriented movements that include 'brain buttons', 'cross crawl' and 'the thinking cap' exercises. Main phase; These are exercises that include coordination, selective attention, audio-visual focus and balance, consisting of perceptual, independent and dependent movements. Cooling phase; It aims to ensure hand-eye coordination by consisting of double doodle, throwing balls to each other and lazy 8s exercises.Exercises were selected from the kinetic brain exercise pool, modified and applied for 2-8 weeks.The exercises were done while sitting and standing, with increasing difficulty levels. The factor that made the levels difficult was the time and complexity of the incoming command. A game ball with a diameter of 7 cm was used for the exercises.
  Arms: Group 1
Other: Core Stabilization Exercises — Core Stabilization Exercise Program in groups of 8-10 people, for 40 minutes, 2 days a week, for 8 weeks.These exercises included a 5-minute active warm-up, a 30-minute Core Stabilization exercise that included upper and lower extremity movements, and immediately followed by a 5-minute cool-down exercise.The exercises are pilates-based and in the first stage of the program. Movements were performed in standing and sitting positions.Movements were started with 6-8 repetitions, increased by 1-2 repetitions each week, and in the last week, 12-15 repetitions were performed, with contraction times increasing from 5 seconds to 10 seconds. As the exercises progressed from easy to difficult, from simple movements to complex movements, the movements were continued by adding an elastic band and 0.5 kg weight.While advancing the exercise program, the exercises were personalized by taking into account the individual's strain levels.

SUMMARY:
The aim of the study is to evaluate the balance and dual-task activities of Kinetic Brain Exercises in healthy elderly individuals living in nursing homes.

DETAILED DESCRIPTION:
A total of 33 people, 4 women and 29 men between the ages of 65-80 (73.88±3.69 years) completed in the research. Demographic and clinic information of the individuals were recorded and Dual Task Performance Tests for dual task activities, Timed Up and Go Test (TUGT) , Functional Reach Test for balance, 10 Meter Walk Test for walking speed, Fall Efficacy Scale (FES) for the fear of falling, Dual Task Questionnaire for to determine individuals difficulties during dual tasks and World Health Organization Quality of Life Instrument- Older Adults Module (WHOQOL-OLD) was used for quality of life. Individuals were applied an exercise program of 40 minutes, 2 days a week for 8 weeks. Individuals were divided into 2 groups. Kinetic Brain Exercises and Core Stabilization Exercises were applied to Group 1 (n=17), and only Core Stabilization Exercises were applied to Group 2 (n=16).

ELIGIBILITY:
Inclusion Criteria:

* Individuals living in nursing homes between the ages of 65-80,
* Having signed the Informed Volunteer Consent Form,
* Sufficient cognitive functions (Mini Mental State Test score being 24 and above)
* Those who can stand independently on their own

Exclusion Criteria:

* Those with neurological, musculoskeletal, inner ear or eye diseases that will cause impairment in vision or standing balance,
* Those with moderate and severe congenital heart disease, coronary heart disease and cerebrovascular disease

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Demographic and Clinical Evaluation Form | At baseline and after 8 weeks
  Name-surname, age, telephone number, gender, education level, height, weight, Body Mass Index (BMI), presence of chronic disease, regular medication use, whether or not they have a hobby, duration of stay in the nursing home, reason for staying in the nursing home and use of assistive walking devices were questioned.
Mini Mental State Test | At baseline and after 8 weeks
  Cognitive status was evaluated.
Dual Task Performance Tests | At baseline and after 8 weeks
  To evaluate dual-task activities, Timed Up and Go Test, 30-Second Sit-and-Go Test, Tandem Stance Test, 360° Rotation Test and One-Leg Stand Test were applied to individuals in three different ways: single task, cognitive task and motor task, and performance times were measured.
10 Meter Walking Test | At baseline and after 8 weeks
  It was used to evaluate individuals' walking speed.
Functional Reaching Test | At baseline and after 8 weeks
  It was used to evaluate the balance performance of individuals.
Dual Task Survey | At baseline and after 8 weeks
  It was used to obtain information about the difficulties individuals experience in daily life situations that require dual tasks.
Tinetti Fall Activity Scale | At baseline and after 8 weeks
  It was used to assess individuals' fear of falling.Minimum score is 0 and maximum score is 28.
World Health Organization Quality of Life Scale Elderly Module | At baseline and after 8 weeks
  It was used to evaluate the quality of life of the elderly. Minimum score is 0 and maximum score is 135.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided